CLINICAL TRIAL: NCT02323386
Title: Anatomo-functional Correlation Between Intra-operative Passive Kinematics Recorded by Navigation and Post-operative Kinematics Analyzed by Dynamic Weight Bearing RSA of the Operated Knee.
Brief Title: Kinematic Analysis of a PS, FB Primary Total Knee Arthroplasty (ATTUNE Knee System) Using Dynamic RSA
Acronym: Attune-RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full professor, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 46/13
Record Dates: First submitted 2014-12-10; First posted 2014-12-23 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis
Keywords: Dynamic RSA; Knee; Total Knee Arthroplasty; Kinematic Analysis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATTUNE knee system (Experimental): The patients will undergo primary Total Knee Arthroplasty (ATTUNE knee system)
  Interventions: Device: Primary Total Knee Arthroplasty (ATTUNE Knee System)

INTERVENTIONS:
Device: Primary Total Knee Arthroplasty (ATTUNE Knee System) — The patient will undergo primary Total Knee ArthroplastY use ATTUNE Knee System. During surgery a navigation system will be used to record preoperative joint kinematics under different tests. During the test the 6 degrees of freedom (DOF) of the joint will be computed and shown to the surgeon; these are the femoral rotation and translation pattern against flexion ranges. Navigation system will be also used to monitor the implant positioning and possible surgical bias. Dynamic RSA will be used to analyze the in vivo kinematics of the prosthesis at 6 months follow-up.
  The above mentioned motion tests will be performed 3 times. The first 2 will be executed to gain comfort with the experimental set-up with no X-ray exposure. During the last data is collected.

SUMMARY:
Background: Across the European Union there are 535,000 Total Knee Arthroplasty (TKA)per year. Statistics indicate that for patients over 60 year old approximately one out of 20 will require corrective reoperations within 10 years after surgery. However, for patients younger than 60 years, approximately one out of 10 will require revision total knee arthroplasty within 10 years of surgery. As the number of younger patients is increasing, there has been a shift in focus in total Knee Replacement (TKR) outcome, with post-operative function and implant longevity being the important issues for quality of patient care. Furthermore, it has been reported that up to 25% of patients are not satisfied with the functional results of their TKA. In vivo the gold standard for obtaining reliable 3D measurements is RSA. However these are often static, because of even most advanced x-ray film exchanger limit the number of pictures taken to less than 10 per second. Our dynamic RSA technique allows producing real time x-ray video of TKA in weight-bearing (WB) conditions with active muscle contraction.

The purpose of this study is to investigate the effect of a new implant design on the post-operative active knee kinematics, focusing on mid-flexion instability of the joint. A prospective randomized study will be performed on a new implant: the DePuy ATTUNETM fixed-bearing (FB) posterior-stabilized (PS) knee prosthesis.

DETAILED DESCRIPTION:
The main goal of this study is to investigate the effect of a new implant design on the postoperative active knee kinematics on mid-flexion instability of the joint. Data will be collected during the surgery with a Computer Assisted Surgery system and in the post operative follow up phase using the dynamic RSA focusing. A prospective study will be performed on a new implant: the DePuy ATTUNETM fixed-bearing (FB) posterior-stabilized (PS) knee prosthesis.

Kinematic tests will be performed to analyze femoral rotation patterns and translation patterns of the medial and femoral condyle respect to the tibial plateau during different daily life motor tasks.

Despite reportedly good implant survival rates, not all patients are fully satisfied after total knee arthroplasty (TKA). One of the most debated topics in TKA is the effectiveness of the prosthesis to reproduce physiological kinematics at the replaced knee, usually expressed in terms of patterns of joint rotation in the three anatomical planes, of the functional axis, and of the tibio-femoral contact points on the medial and lateral condyles, that is, femoral roll-back.

Implant design can influence final kinematic results. The mid-flexion instability may be the cause of joint instability, paradoxical femoral rollback, surgical variation.

Recently an improved implant design of fixed bearing PS DePuy implant has been anticipated to early users. This implant has been claimed to reduce midflexion instability and improve joint kinematics, because of a particular multiradius shape of the condylar surface.

For intra-operative kinematic acquisition, a commercial navigation system (BLUIGS, Orthokey Italia srl, Firenze, Italy) with a dedicated software for kinematic tests will be used.

In the present study, the investigators will use a postoperative bi-planar imaging method in weight-bearing motor tasks with active muscle contraction , to determine the in vivo contact areas on the tibial articulating surface of a PS TKA during flexion of the knee.

The objective of the present study is to determine the contact areas and their movement through a 0-140° arc of motion in both the anteroposterior (AP) and ML directions. The cohort will also be compared with data of normal knee kinematics, as reported in current literature.

At 6 months follow-up, dynamic fluoroscopy will be used to analyze implant kinematics (i.e. stair descent, level-walking and non weight-bearing maximum knee flexion) and a simultaneous, real-time collection of ground reaction forces with a force platform will be performed. Clinical scores will be collected at that time and compared with all the data registered before surgery and during the follow up routinely made at 1 and 3 months after surgery.

A specifically developed device installed at the Rizzoli Orthopaedic Institute will be used to assess the kinematic of the knee at 9 months after surgery. This equipment is unique worldwide: it was specifically designed, built and certified for dynamic and static RSA evaluation of TKA. The purpose of this study is to investigate the effect of a new implant design on the post-operative active knee kinematics, focusing on mid-flexion instability of the joint. A prospective randomized study will be performed on a new implant: the DePuy ATTUNETM fixed-bearing (FB) posterior-stabilized (PS) knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Severe radiographic osteoarthritis (Kellgren-Lawrence grade >3)
* Patients scheduled for a primary TKA
* Willing to take part in study and providing HIPAA authorization

Exclusion Criteria:

* Previous corrective osteotomy on the affected lower limb
* Post-traumatic arthritis
* Severe preoperative valgus deformity (Hip Knee Ankle angle>10°)
* BMI>40 kg/m2
* Rheumatoid arthritis
* Chronic inflammatory joint diseases
* Patients with a pre-pathological abnormal gait (amputated, neuromuscular disorders, poliomyelitis, developmental dysplasia of the hip)
* Severe ankle osteoarthritis (Kellgren-Lawrence>3)
* Severe hip osteoarthritis (Kellgren-Lawrence>3)
* Previous total hip or ankle replacement
* Unwilling to take part in study and providing HIPAA authorization

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the femoral rotations and translations during weight-bearing motor tasks with active muscle contraction: step descent, full flexion movement, level walking. | 9 months
  The joint kinematic was acquired using the dynamic RSA technique. The rotations (angular degree) and translations (millimeter) were evaluated using the Euler decomposition and the Low-point algorithm.

SECONDARY OUTCOMES:
Correlation of clinical reported results (KSS, Oxford, SF36, WOMAC) and patients' subjective satisfaction using a visual analogue scale (VAS) with kinematics differences and ground reaction forces. | 9 months
  KSS, OXFORD, SF36, WOMAC, VAS scores will be assessed and recorded pre-operatively and post operatively at 6 months after surgery
Quantification the ground reaction forces during weight-bearing motor tasks with active muscle contraction: step descent, full flexion movement, level walking. | 9 months
  Forces (newton N)

CONTACTS AND LOCATIONS:
Overall Officials: Maurilio Marcacci, MD, Principal Investigator — Rizzoli Orthopaedic Institute; Laura Bragonzoni, SportScience, Study Director — Alma Mater Studiorum - University of Bologna; Danilo Danilo, MD, Study Chair — Rizzoli Orthopaedic Institute; Bontempi Marco, Physicist, Study Director — Rizzoli Orthopaedic Institute; Maria Pia Neri, MD, Study Chair — Rizzoli Orthopaedic Institute
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
The IPd are to be shared by papers

REFERENCES:
- [Derived] Di Paolo S, Agostinone P, Grassi A, Lucidi GA, Pinelli E, Bontempi M, Marchiori G, Bragonzoni L, Zaffagnini S. Dynamic Radiostereometry Evaluation of 2 Different Anterior Cruciate Ligament Reconstruction Techniques During a Single-Leg Squat. Orthop J Sports Med. 2021 Jul 15;9(7):23259671211011940. doi: 10.1177/23259671211011940. eCollection 2021 Jul. PMID 34350300